CLINICAL TRIAL: NCT02739737
Title: Testing for the Presence of Authorship Bias in Peer Review
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Seth Leopold, Professor, Dept of Orthpaedics and Sports Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 46129-EA
Record Dates: First submitted 2016-04-04; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Peer Review
Keywords: Bias; Orthopedics; Peer Review

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blinded Reviewers (Experimental): Subjects receiving randomized sham manuscript for review
  Interventions: Other: Blinded manuscript
- Unblinded Reviewers (Experimental): Subjects receiving randomized sham manuscript for review
  Interventions: Other: Unblinded manuscript

INTERVENTIONS:
Other: Blinded manuscript — Blinded version of sham manuscript
  Arms: Blinded Reviewers
Other: Unblinded manuscript — Unblinded version of sham manuscript
  Arms: Unblinded Reviewers

SUMMARY:
No consensus exists among biomedical journals on the subject of blinding during the peer review process. Some journals attempt to remove all identifiers of authorship from potential manuscripts before delivering to referees for peer review while others prefer to leave the authorship transparent. Although peer review remains the gold standard for manuscript evaluation, the lack of a standardized blinding process between editorial offices may be a source of publication bias and make comparisons of manuscripts published in different journals more difficult to interpret.

Proponents of a blinded peer review system believe that knowledge of authorship may leave referees vulnerable to biases about those authors' previous research, perceived expertise, institution, nationality, or gender. This shifts judgment away from the merits of the scientific work and introduces pre-conceived notions about the identity and background of the author into the review process. Conversely, supporters of transparent authorship argue that knowledge of author identity makes it easier for the referee to provide more appropriate critiques. Open author identification allows referees to compare the current manuscript to previously published work by the author, and to recognize or identify potentially important conflicts of interest.

The investigators therefore propose an experimental study to address the question of whether blinding affects the likelihood a reviewer will recommend acceptance of a study being peer reviewed. The investigators plan to work in partnership with a journal to have a fabricated manuscript peer reviewed by a large number of reviewers; the authors will send this "test" manuscript out either in blinded form (authors' names/institutions not shown to reviewers) or in open form, with the names of several well-known, well-regarded authors and their institutions visible to peer reviewers. The manuscripts will otherwise be identical.

The partnering journal, Clinical Orthopaedics and Related Research allows both open and blinded peer review, regularly employing both approaches (authors can choose what kind of review they prefer when they submit to CORR), and so the reviewers are unlikely to be troubled by seeing a manuscript in either format.

The primary goal of this study is to determine whether the identification of a manuscript with a prominent group of authors (open authorship) will affect the likelihood that reviewers will recommend the manuscript for publication.

Additionally, the investigators plan to purposely place several errors in the manuscript, and tally how often reviewers detect these mistakes, to determine whether reviewers read the work of prominent authors less critically.

The investigators will also compare the reviewers' grading of the (identical) methods section, to determine whether the identification of a manuscript with prominent authors results in higher reviewer grades for methodological rigor.

This study tests the following specific hypotheses:

1. The visibility of prominent author names and institutions on test manuscripts will be associated with increased likelihood that the manuscript will be recommended for publication by peer reviewers. (Primary Study Endpoint)
2. The visibility of prominent author names and institutions will be associated with a decreased likelihood that purposefully placed "errors" in the experimental manuscript will be detected by the reviewers.
3. The visibility of prominent author names and institutions will be associated with increased scores given by reviewers for the methods section, despite the fact that the methods sections of the experimental manuscript will be identical.

NOTE:

All elements of the research protocol were approved by the University of Washington Human Subjects Review Committee, including the study's opt-out design for reviewer recruitment, since it was considered important that reviewers not know that the paper they evaluated was part of a study. To minimize the potential for harm, the authors chose as the topic of the fabricated test manuscript an intervention that could not be immediately put into practice at reviewers' own centers (a particular team-training process in the operating room). In addition, participating reviewers were informed which paper was the test manuscript at the completion of data collection, so that they did not pursue this sort of team training based on the results of the fabricated study.

To reduce the risk of an observer (Hawthorne) effect, it was important to minimize the likelihood that participant reviewers would learn of the study while it was in progress. To this end, the investigators elected not to pre-register the study in a trial registry.

ELIGIBILITY:
Inclusion Criteria:

* Registered peer reviewers in relevant subspecialty sections of CORR's reviewer database.

Exclusion Criteria:

* Reviewers who opt out (electronically, by phone, or by post).

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Manuscript acceptance rate | 13 months

SECONDARY OUTCOMES:
Error detection rate | 13 months
Methods section score | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Seth L Leopold, MD, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Rooyen S, Godlee F, Evans S, Black N, Smith R. Effect of open peer review on quality of reviews and on reviewers' recommendations: a randomised trial. BMJ. 1999 Jan 2;318(7175):23-7. doi: 10.1136/bmj.318.7175.23. PMID 9872878
- [Background] McNutt RA, Evans AT, Fletcher RH, Fletcher SW. The effects of blinding on the quality of peer review. A randomized trial. JAMA. 1990 Mar 9;263(10):1371-6. PMID 2304216
- [Background] Justice AC, Cho MK, Winker MA, Berlin JA, Rennie D. Does masking author identity improve peer review quality? A randomized controlled trial. PEER Investigators. JAMA. 1998 Jul 15;280(3):240-2. doi: 10.1001/jama.280.3.240. PMID 9676668
- [Background] Fisher M, Friedman SB, Strauss B. The effects of blinding on acceptance of research papers by peer review. JAMA. 1994 Jul 13;272(2):143-6. PMID 8015127
- [Background] Emerson GB, Warme WJ, Wolf FM, Heckman JD, Brand RA, Leopold SS. Testing for the presence of positive-outcome bias in peer review: a randomized controlled trial. Arch Intern Med. 2010 Nov 22;170(21):1934-9. doi: 10.1001/archinternmed.2010.406. PMID 21098355
- [Derived] Okike K, Hug KT, Kocher MS, Leopold SS. Single-blind vs Double-blind Peer Review in the Setting of Author Prestige. JAMA. 2016 Sep 27;316(12):1315-6. doi: 10.1001/jama.2016.11014. No abstract available. PMID 27673310